CLINICAL TRIAL: NCT04641013
Title: Age-related Clonal Haematopoiesis in an HIV Evaluation Cohort (ARCHIVE): a follow-on Study of the Australian Positive & Peers Longevity Evaluation Study
Brief Title: Age-related Clonal Haematopoiesis in an HIV Evaluation Cohort (ARCHIVE)
Acronym: ARCHIVE
Status: Active, not recruiting | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Peter MacCallum Cancer Centre, Australia (Other); Holdsworth House Medical Centre (Unknown); Prahran Market Clinic (Unknown); East Sydney Doctors (Unknown); RPA Sexual Health (Unknown); The Alfred (Other); St Vincent's Hospital (Other); Taylor Square Medical Practice (Unknown); Monash Health (Other); Albion Street Clinic (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-11-ARCHIVE
Record Dates: First submitted 2020-11-12; First posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; Aging
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with HIV over the age of 55 years
- People without HIV over the age of 55 years

SUMMARY:
The ARCHIVE study is an observational longitudinal cohort study of people with and without HIV who are over the age of 55. The duration of the study is planned for 10 years, with study visits every 1-2 years. The objectives of the study are to evaluate genomic and other factors associated with aging, stratified by HIV status.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >55
* For participants without HIV: an HIV negative test within 12 months prior to enrolment. If no HIV-negative test result is available within 12 months prior to enrolment, then participants will be tested for HIV as part of standard of care, if indicated by the guidelines for HIV testing published by the Australasian Society for HIV, Viral Hepatitis and Sexual Health Medicine14. This study will not conduct HIV testing; therefore, any participants without HIV being considered for participation in the study will need to have had a standard of care HIV negative test within the past 12 months. Some subjects at on-going risk for HIV are recommended to have periodic HIV testing and may be due for such testing as part of standard of care, at the time of enrolment into the study.
* Willing and able to provide written informed consent and willingness to participate in and comply with a longitudinal cohort study including 1) consent to providing blood samples for full blood count, inflammatory marker testing and genomics analysis 2) consent to linking their data to national and state-wide data registries (including consent to providing personally identifying information); and 3) consent to participate in future follow-up studies

Exclusion Criteria:

- Unwilling or unable to provide consent to participate

Age Groups: Child, Adult, Older Adult
Study Population: People over the age of 55, with and without HIV
Sampling Method: Non-Probability Sample
Enrollment: 446 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2019-04-17 (Actual); Study Completion 2027-12-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with at least one somatic mutation associated with clonal haematopoiesis | 2017-2019
  Detection of mutations associated with clonal haematopoiesis

SECONDARY OUTCOMES:
Median and natural log-transformed Interleukin-6 | 2017-2019
  Interleukin-6 level
Median (IQR) and natural log-transformed C-reactive protein and Cystatin C; D-dimer >0.27 | 2017-2019
  C-reactive protein, Cystatin C, D-dimer
Median (IQR) and natural log-transformed Haemoglobin | 2017-2019
  Haemoglobin
Median (IQR) and natural log-transformed White blood cell count, Median (IQR) and natural log-transformed Neutrophil count, natural log-transformed Lymphocyte count, natural log-transformed platelet count | 2017-2019
  White blood cell count, Neutrophil count, Lymphocyte count, platelet count
natural log-transformed Mean corpuscular volume | 2017-2019
  mean corpuscular volume
natural log transformed Red Cell distribution width | 2017-2019
  red cell distribution width
Proportion of participants with diagnosed cardiovascular conditions, any malignancy, haematologic malignancies | 2017-2019
  Comorbid conditions

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polizzotto, MBBS, PhD, Principal Investigator — Kirby Institute, UNSW Sydney; Nila Dharan, MD, Principal Investigator — Kirby Institute, UNSW Sydney; Kathy Petoumenos, PhD, Principal Investigator — Kirby Institute, UNSW Sydney
Locations (11):
- Australia (11):
  - St Vincent's Hospital HIV, Immunology and Infectious Disease Unit, Darlinghurst, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - East Sydney Doctors, Sydney, New South Wales
  - Holdsworth House Medical Practice, Sydney, New South Wales
  - Kirby Institute, Sydney, New South Wales
  - Taylor Square Private Clinic, Sydney, New South Wales
  - RPA Sexual Health, Royal Prince Alfred Hospital, Camperdown, Sydney, New South Wales
  - Alfred Hospital, Melbourne, Victoria
  - Prahran Market Clinic, Melbourne, Victoria
  - Monash Medical Centre, Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dharan NJ, Yeh P, Bloch M, Yeung MM, Baker D, Guinto J, Roth N, Ftouni S, Ognenovska K, Smith D, Hoy JF, Woolley I, Pell C, Templeton DJ, Fraser N, Rose N, Hutchinson J, Petoumenos K, Dawson SJ, Polizzotto MN, Dawson MA; ARCHIVE Study Group. HIV is associated with an increased risk of age-related clonal hematopoiesis among older adults. Nat Med. 2021 Jun;27(6):1006-1011. doi: 10.1038/s41591-021-01357-y. Epub 2021 Jun 7. PMID 34099923